CLINICAL TRIAL: NCT04395300
Title: Sleep Quality and Effect on General Health in Healthcare Personnel During COVID-19 Pandemic
Brief Title: Sleep Quality in Healthcare Personnel During COVID-19
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU14
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Sleep Quality; General Health
Keywords: COVID-19; corona virus disease; Pittsburgh sleep quality index; General health questionnare; Healthcare worker
MeSH Terms: conditions — COVID-19; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Physicians, Nurses, Laboratory workers, radiology technicians
  Interventions: Other: Web Based Survey

INTERVENTIONS:
Other: Web Based Survey — On line survey distributed electronically

SUMMARY:
Coronavirus disease 2019 (COVID-19), represents a medical and psychological challenge to healthcare workers to the limits that it affects their quality of sleep and their general health.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare personnel actively working during the pandemic

Exclusion Criteria:

* non healthcare workers

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: physicians, nurses, laboratory and radiology technicians
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
measure sleep quality in healthcare worker | one month
  Pittsburgh sleep quality index (0-21) higher means worse quality

SECONDARY OUTCOMES:
impact of covid-19 pandemic on general health | 40 days
  general health questionnaire (0-12) higher means worse
correlate between sleep quality and general health | 40 days
  web based survey

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No